CLINICAL TRIAL: NCT05089240
Title: Data Collection of Objective Parameters and Subjective Feedback on Visually Fatigued Subjects and Evaluation of the Effect of Ophthalmic Lenses to Alleviate Visual Fatigue
Brief Title: Objective and Subjective Evaluation of Ophthalmic Lenses With Extra Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Collaborators: Elite School of Optometry and Sankara Nethralaya (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ESS-TEC 191
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Asthenopia
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20-29 years (+0.40D extra power) (Other)
  Interventions: Device: Ophthalmic lens with extra power
- 30-35 years (+0.40D extra power) (Other)
  Interventions: Device: Ophthalmic lens with extra power
- 20-29 years (+0.40D extra power with blue cut) (Other)
  Interventions: Device: Ophthalmic lens with extra power

INTERVENTIONS:
Device: Ophthalmic lens with extra power

SUMMARY:
To evaluate subjective visual performance and objective visual parameters when wearing ophthalmic lenses with extra power (+0.4 D or +0.6 D), and ophthalmic lenses with a selective blue cut filter.

ELIGIBILITY:
Inclusion Criteria:

* Subjective report of visual fatigue
* Non-presbyopes
* Permanent wearers who wear glasses for at least 5 hours a day
* Distance refractive error within the range of [+6.00 to -6.00]* (with cylinder in the negative form),
* Cylindrical component of the refractive error within the range of 0 to 2 D in both eyes,
* Anisometropia ≤ 1.00 D in sperical equivalent,
* Visual acuity of +0.10 logMAR or better in each eye with new prescription at distance (high contrast/high luminance),
* Distance visual acuity difference ≤0.20 logMAR between right and left eye (high contrast, high luminance)
* Near binocular visual acuity of +0.10 logMAR or better with a new prescription (high contrast, high luminance),
* Study frame characteristics: Frame B size at least 22 mm

Exclusion Criteria:

* Vulnerability of the subject,
* Participation in another study which might have an influence on vision or interfere with study assessments,
* Binocular vision problems,
* Known ocular pathology (e.g., age-related macular degeneration, glaucoma…),
* Any previous ocular surgery which might have an influence on vision or interfere with study assessments (e.g., iridectomy, refractive surgery…),
* Any untreated and/or uncontrolled systemic condition which might have an influence on vision, or interfere with study assessments (e.g., uncontrolled diabetes, uncontrolled high blood pressure…),
* Any medical treatment or medication that might have an influence on vision or interfere with study assessments (e.g., antidepressants, drugs with atropinic effects…),
* Knowledge/expertise in optometry, ophthalmic lenses, or optics based on past or current professional activity (e.g., optometrists, opticians, ophthalmologists…)

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
The difference in number of participants with treatment-related adverse events between the two lenses | Immediately after the first and second wearing period (21 days each)
  Any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device. Determined by subject's spontaneous reporting, the Investigator's non-leading questioning and his/her evaluation.